CLINICAL TRIAL: NCT04695119
Title: Sepsis in the Intensive Care Unit-II
Brief Title: Sepsis in the ICU-II
Status: Recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Ryhov Hospital, Jönköping (Unknown); Bicetre Hospital (Other); HÃ´pital EuropÃ©en George Pompidou, APHP, Paris, France (Unknown)
Responsible Party: Principal Investigator, Michelle Chew, Professor, Linkoeping University
Other Study IDs: SICU-II
Record Dates: First submitted 2020-12-21; First posted 2021-01-05 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Septic Shock; Sepsis; Cardiomyopathies; Organ Failure, Multiple
MeSH Terms: conditions — Shock, Septic; Sepsis; Cardiomyopathies; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma isolated neutrophils bronchoalveolar lavage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients with septic shock: All adult (>=18 yo) patients admitted to participating ICUs with septic shock defined according to the Sepsis III criteria.
  Purely observation study with no intervention. Patients are exposed to septic shock and treatment according to standard departmental protocols at each centre.
  Interventions: Other: Exposure is septic shock (defined according to Sepsis-III) and standard treatment according to departmental protocols.

INTERVENTIONS:
Other: Exposure is septic shock (defined according to Sepsis-III) and standard treatment according to departmental protocols. — Collection of data, biomarker and echocardiography analysis will be centralized and blinded. Assessment of endpoints will be blinded.

SUMMARY:
Sepsis-induced cardiac dysfunction (SIMD) is a well-known phenomenon yet its diagnosis remains elusive with no accepted definition, or defining pathophysiological mechanism associated with this disease. Systolic dysfunction occurs in 20-70% of patients, and may be severe, yet does not appear to have any prognostic value for mortality. Diastolic function has also been variably described and seems to be related to short-term mortality. However, the contribution of left ventricular systolic and diastolic dysfunction to mortality in sepsis are still far from clear, with uncertain contribution from previous cardiovascular disease, vasopressor and inotropic drugs and mechanical ventilation. Another poorly investigated area is right ventricular dysfunction. Cor pulmonale occurs in up to 25% of patients with septic shock, and is invariably related to pulmonary haemodynamics and mechanical ventilation, yet very little is known about how this affects prognosis. Finally, although the outcome of disease is a function of multiple parameters, septic cardiomyopathy is most frequently characterized based on individual echocardiographic parameters, without considering their interactions or placing them in the context of biomarkers and clinically available haemodynamic data. Available relevant studies are often monocentric, and many fail to consider the various confounders that influence the clinical outcome in sepsis. Therefore, the diagnostic and prognostic value of combinations of clinical, biochemical and haemodynamic variables remains to be established.

Accordingly, the purpose of this study is to identify biomarkers and echocardiographic and haemodynamic signatures characteristic of specific outcomes in SIMD to support the diagnosis and prognosis in SIMD. Specific aims are:

1. To determine the association between left ventricular systolic and diastolic dysfunction, and adverse outcome in SIMD;
2. To determine the association between right ventricular systolic and diastolic dysfunction, and adverse outcome in SIMD;
3. To determine the association between novel biomarkers and adverse outcome in SIMD;
4. To determine the combined value of biomarker, echocardiographic, and haemodynamic variables for predicting adverse outcomes in SIMD;
5. To explore if there are different phenotypes of SIMD using unsupervised machine learning algorithms, and whether they are associated with adverse outcomes.

50 patients will be enrolled in a feasibility study to evaluate the logistical setup for acute echocardiography and biobanking facilities. A further 300 patients will be enrolled with inclusion from peripheral centers once feasibility is confirmed.

DETAILED DESCRIPTION:
UPDATE 26 Feb 2022:

A pilot project was completedafter recruitment of 50 patients confirming the feasibility of data collection, study logistics, biomarker assay set-up and frequency of outcomes. Cancellation of non-COVID related research in 2020&2021 has caused significant delays. Recruitment of patients will continue during 2022&2023. At the time of writing 70 patients have been recruited across 4 centres.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to ICU and fulfilling the Sepsis-III criteria for septic shock

Exclusion Criteria:

* No informed consent
* Acute coronary syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to participating ICUs with a presumptive diagnosis of septic shock will be screened for eligibility. Patients fulfilling the Sepsis-III criteria for septic shock will included. Study inclusion must occur within 12h of ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury | any time during ICU stay within the study period, up to 10 days
  increased hsTnT
Organ failure free days | 30 days of study inclusion
  Organ failure

SECONDARY OUTCOMES:
30 day mortality | 30 days after study inclusion
  Short term mortality
365 day mortality | 365 days after study inclusion
  Long term mortality

OTHER OUTCOMES:
Exploratory outcomes | during ICU stay, up to 10 days
  Vasopressor inotropic score
Exploratory outcomes | 30 days of study inclusion
  Days free of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chew, MBBS, PhD, Study Chair — Linkoeping University Hospital; Bernard Cholley, MD, PhD, Principal Investigator — CHU George Pompidou; Belaid Bouhemad, MD, PhD, Principal Investigator — CHU Dijon; Fredrik Hammarsköjld, MD, PhD, Principal Investigator — Ryhov Hospital, Jönköping; Xavier Monnet, MD, PhD, Principal Investigator — Hopital Bicetre
Locations (4):
- France (2):
  - CHU Dijon-Bourgogne, Dijon, Dijon
  - CHU Georges Pompidou, Paris, Paris
- Sweden (2):
  - Ryhov Sjukhus Jönköping, Jönköping, Jönköping County
  - Dept of Anaesthesia and Intensive Care, Linköping

REFERENCES:
- [Derived] Blixt PJ, Nguyen M, Cholley B, Hammarskjold F, Toiron A, Bouhemad B, Lee S, De Geer L, Andersson H, Aneq MA, Engvall J, Chew MS. Association between left ventricular systolic function parameters and myocardial injury, organ failure and mortality in patients with septic shock. Ann Intensive Care. 2024 Jan 18;14(1):12. doi: 10.1186/s13613-023-01235-5. PMID 38236316